CLINICAL TRIAL: NCT01424163
Title: A Single and Multiple Dose, Open-Label Study of the Pharmacokinetics, Safety, and Tolerability of Dexpramipexole (BIIB050) in Healthy Japanese and Caucasian Subjects
Brief Title: Dexpramipexole Japanese PK Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Knopp Biosciences (Industry)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 223HV101
Record Dates: First submitted 2011-07-28; First posted 2011-08-26 (Estimated); Last update posted 2021-06-22 (Actual); Status verified 2014-11

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment 1 (Part A) (Experimental): Dexpramipexole single dose (reduced dose)
  Interventions: Drug: Single dose reduced
- Treatment 2 (Part A) (Experimental): Dexpramipexole single dose (Standard dose)
  Interventions: Drug: Single dose standard
- Treatment 3 (Part A) (Experimental): Dexpramipexole multiple dosing
  Interventions: Drug: Multiple Dose
- Treatment for Part B (Experimental): Dexpramipexole multiple dosing
  Interventions: Drug: Multiple Dose

INTERVENTIONS:
Drug: Single dose reduced — Treatment 1 (Part A)
  Arms: Treatment 1 (Part A)
Drug: Single dose standard — Treatment 2 (Part A)
  Arms: Treatment 2 (Part A)
Drug: Multiple Dose — Treatment 3 (Part A)
  Arms: Treatment 3 (Part A)
Drug: Multiple Dose — Part B
  Arms: Treatment for Part B

SUMMARY:
This is a single and multiple dose, open-label study to evaluate the pharmacokinetics (PK), safety, and tolerability of dexpramipexole administered orally to adult Japanese and Caucasian healthy subjects.

DETAILED DESCRIPTION:
The study is designed to evaluate the influence of ethnic factors on dexpramipexole safety, tolerability, and PK. Subjects will be admitted to the clinical unit on Day -1 (the day prior to first dosing) and will remain in the clinical unit under observation until discharge. All subjects will have a final follow up visit. Whilst resident in the clinic, subjects will receive 4 treatments: The first 3 treatments comprise Part A of the study and the final treatment group comprises Part B.

Part A:

Treatment 1: Dose 1 (reduced) of dexpramipexole; a single dose Treatment 2: Dose 2 (standard) dexpramipexole; a single dose Treatment 3: Dose 3 (standard) dexpramipexole; 5 doses administered at 12 hour intervals Part B: Dose 4 (standard) dexpramipexole; 5 doses administered at 12 hour intervals There will be a minimum washout of 3 days between treatments.

For all subjects, prior to proceeding to the next treatment group, safety and tolerability data will be reviewed.

Caucasian subjects will be matched individually (on a 1:1 basis) to Japanese subjects with respect to gender and age and if possible BMI.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are able and willing to give written informed consent.
* Adult Japanese and Caucasian males/females aged 18 to 60 years inclusive and between 18 and 30 kg/m2 body mass index (BMI), inclusive.
* Male and female subjects will be enrolled on the study. Male subjects and female subjects of childbearing potential, must practice effective contraception during the study and be willing and able to continue contraception for 1 month (females) or 3 months (males) after their last dose of study treatment
* Japanese subjects must be born in Japan and have both parents and four grandparents of Japanese descent.
* Japanese subjects must have lived outside of Japan for no more than 5 years.
* Japanese subjects must not have significant changes with regard to diet; i.e., their diet must not have significantly changed since leaving Japan.
* Caucasian subjects will be matched individually (on a 1:1 basis) to Japanese subjects with respect to gender and age, and if possible BMI.

Exclusion Criteria:

* Subjects who do not conform to the above inclusion criteria.
* Female subjects who are pregnant, trying to become pregnant or lactating.
* Subjects who have a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases or disorders.
* Subjects who have a clinically relevant surgical history.
* Subjects who have previously received dexpramipexole or pramipexole.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2011-08; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Cmax of dexpramipexole | pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours after dosing on Days 1 and 5 in Treatments 1 and 2, and after the fifth dose on Day 11 in Treatment 3 for Parts A & B.
AUC of dexpramipexole | pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours after dosing on Days 1 and 5 in Treatments 1 and 2, and after the fifth dose on Day 11 in Treatment 3 for Parts A & B.

SECONDARY OUTCOMES:
Changes in clinical laboratory tests | pre-dose to 72 hrs post-dose in each dose group and again at follow-up (14 hrs post last dose)
ECG changes | pre-dose to 72 hrs post-dose in each dose group and again at follow-up (14 hrs post last dose)
Vital Sign changes | pre-dose to 72 hrs post-dose in each dose group and again at follow-up (14 hrs post last dose)
Adverse Event monitoring | pre-dose to 72 hrs post-dose in each dose group and again at follow-up (14 hrs post last dose)

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, London, United Kingdom